CLINICAL TRIAL: NCT00821613
Title: Collection of Raw Data of Thermal Imaging for the Purpose of Developing a Device for Early Detection of Breast Cancer
Brief Title: Data Collection Study of Raw Thermal Images for the Purpose of Developing a Device for Early Detection of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Real Imaging Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: Pr-118-8061 ver. 004; QMS number: 960-PRL-09011
Record Dates: First submitted 2009-01-12; First posted 2009-01-13 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only
Oversight: Data Monitoring Committee: No

SUMMARY:
Collection of thermal "images" of women with breast tumors in varying degrees of severity and of healthy women with no breast findings, in order to evaluate and improve Real Imaging's device ("RI4.0"), capabilities which will assist in early detection of breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Gender: female
* Age: 18 years and older
* Subjects with a breast abnormality (identified by mammography, ultrasound, MRI and/or a clinical examination) summoned for breast biopsy or subjects summoned for a routine screening examination.
* Subject who have signed an informed consent form.

Exclusion Criteria:

* Subjects who have had a mammography, ultrasound, and/or MRI examination performed on the day of the study, prior to being "imaged" by RI4.0.
* Subjects who have undergone any type of breast surgery throughout the 6 weeks preceding the study.
* Subjects who have had a breast biopsy performed throughout the 6 weeks preceding the study.
* Subjects who have undergone a mastectomy.
* Subjects who have a large scar (causing breast deformation) following breast lumpectomy and/or any other cause (e.g. accident).
* Subjects with prior breast reduction surgery or breast augmentation surgery.
* Subjects who have a fever on the day of their biopsy.
* Subjects who are pregnant.
* Subjects who are breast-feeding.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects with a breast abnormality (identified by mammography, ultrasound, MRI and/or a clinical examination) summoned for breast biopsy or subjects summoned for a routine screening examination.
Sampling Method: Non-Probability Sample
Enrollment: 1827 (Actual)
Dates: Start 2009-09; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- Israel (6):
  - Hadassah Ein Kerem Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
  - Assuta Ramat Hachayal Hospital, Tel Aviv